CLINICAL TRIAL: NCT02839473
Title: Hydrosorb® Versus Control (Water Based Spray) in the Management of Radio-induced Skin Toxicity: Multicentre Controlled Phase III Randomized Trial
Brief Title: Hydrosorb® Versus Control in the Management of Radio-induced Skin Toxicity: Multicentre Controlled Phase III Randomized Trial
Acronym: HYDROSORB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Paul Hartmann (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2009-07
Record Dates: First submitted 2016-07-08; First posted 2016-07-21 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Radiation Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrosorb® arm (Experimental): Hydrogel Hydrosorb®
  Interventions: Device: Hydrogel Hydrosorb®
- Placebo arm (Placebo Comparator): Castalie water spray
  Interventions: Device: Castalie water spray

INTERVENTIONS:
Device: Castalie water spray
  Arms: Placebo arm
Device: Hydrogel Hydrosorb®
  Arms: Hydrosorb® arm

SUMMARY:
The primary objective consisted of avoiding deterioration and/or restoring the integrity of the skin of patients treated by radiotherapy, right from the first signs of grade 1 or 2 radiation dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Women treated by normo fractionated radiotherapy for breast cancer
* Presenting grade 1 or 2 radiation dermatitis during the treatment and who provided their written informed consent were included in the study.

Exclusion criteria:

* Were male patients
* Radiation dermatitis already treated or caused by another treatment
* Subjects deprived of their freedom or under guardianship
* Subjects in whom medical follow-up was impossible
* A cancer wound or skin flap on the irradiated zone
* A history of allergic skin reaction
* Concomitant chemotherapy or concomitant bevacizumab therapy and bilateral irradiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
local treatment failure defined as interruption of radiotherapy because of skin radiotoxicity or change of local care because skin alteration. | through study completion, an average of 3 years

SECONDARY OUTCOMES:
skin colorimetry measured by a colorimeter | day0, day 7, day 14, day 21, day 28
pain level assessed by the visual analog pain scale | day0, day 7, day 14, day 21, day 28
quality of life assessed with the Dermatology Life Quality Index questionnaire | day0, day 14, day 28

CONTACTS AND LOCATIONS:
Overall Officials: Youlia Kirova, MD, Principal Investigator — Institut Curie
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Centre René Huguenin, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Bazire L, Fromantin I, Diallo A, de la Lande B, Pernin V, Dendale R, Fourquet A, Savignoni A, Kirova YM. Hydrosorb(R) versus control (water based spray) in the management of radio-induced skin toxicity: Results of multicentre controlled randomized trial. Radiother Oncol. 2015 Nov;117(2):229-33. doi: 10.1016/j.radonc.2015.08.028. Epub 2015 Aug 29. PMID 26328937